CLINICAL TRIAL: NCT04393064
Title: Fiberoptic Endoscopic Evaluation of Swallowing(FEES) in Infants Graduated From (NICU) Neonatal Intensive Care Unite
Acronym: FEES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Lamiaa Mohamed Abdel Motaleb, Neonatal specialist, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FEES IN INFANTS
Record Dates: First submitted 2020-04-09; First posted 2020-05-19 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Fiberoptic Endoscope Evaluation of Swallowing in Infants(FEES)

STUDY DESIGN:
Intervention Model Description: 75 preterm and 75 fullterm will be recruited in this study; all will be hemodynamically stable on discharge then doing FEES
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- full term and preterm (Other): 75 preterm and 75 fullterm will be recruited in this study; all will be hemodynamically stable on discharge doing FEES
  Interventions: Device: fiberoptic endoscopic evaluation of swallowing

INTERVENTIONS:
Device: fiberoptic endoscopic evaluation of swallowing — intreventions name :-Fiberoptic endoscopic evaluation of swallowing(FEES) will be performed on all infants enrolled in this study.
  interventions type: flexible nasopharyngeal laryngoscope 3,5 mm in size with portable camera & light source & video recording system will be used. Procedure will be done without anesthesia
  .

SUMMARY:
Based on study showing the ability of using FEES in infant in NICU; so the aim of this study to screen the newborns graduated from NICU using clinical bed side evaluation as well as flexible endoscopic assessment of swallowing to identify the ones suffering from oropharyngeal and / or esophageal dysphagia as well as newborns at risk for aspiration &aspiration pneumonia to tailor or identify appropriate feeding plan for those high risk popularities and support them

DETAILED DESCRIPTION:
* Population study& disease condition Newborns that are discharged from NICU and are hemodynamically stable.
* Interventions The following study will be conducted in neonatal intensive care unit of Kasr alany and Abu EI-Rish hospital, also conducted in Phoniatrics Outpatient of Kasr alany, Cairo university This study will recruit 75 preterm and 75 fullterm will be recruited in this study; all will be hemodynamically stable on discharge

ELIGIBILITY:
Inclusion Criteria:

* Item

  * Neonates who discharged from NICU as they are hemodynamic stable

Exclusion Criteria:

* Item

  * Neonates with congenital anomalies that interfere with the introduction or the procedure of FEES as nasal deformities, choanal atresia, cleft lip and cleft palate.
  * Neonates have liver disease and/ or bleeding tendency

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Fiberoptic endoscopic evaluation of swallowing (FEES) | baseline
  to identify the ones suffering from oropharyngeal and / or esophageal dysphagia as well as newborns at risk for aspiration &aspiration pneumonia by FEES to tailor or identify appropriate feeding plan for those high risk popularities and support them

SECONDARY OUTCOMES:
Other imaging procedures including X-ray (Chest & abdominal) , U/S(ultrasound) , CT(computer tomography) & ECHO(Echocardiography) | baseline
  for any disorder affecting swallowing

CONTACTS AND LOCATIONS:
Overall Officials: Dina Akmal, MD, Study Director — assistant professour; Engy Tosson, MD, Study Director — assistant professour; Ayaallah Shekhany, MD, Study Director — assistant professour
Locations (1):
- Lamiaa Mohamed, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Willette S, Molinaro LH, Thompson DM, Schroeder JW Jr. Fiberoptic examination of swallowing in the breastfeeding infant. Laryngoscope. 2016 Jul;126(7):1681-6. doi: 10.1002/lary.25641. Epub 2015 Sep 15. PMID 26372024
- [Background] da Silva AP, Lubianca Neto JF, Santoro PP. Comparison between videofluoroscopy and endoscopic evaluation of swallowing for the diagnosis of dysphagia in children. Otolaryngol Head Neck Surg. 2010 Aug;143(2):204-9. doi: 10.1016/j.otohns.2010.03.027. PMID 20647120
- [Background] Sitton M, Arvedson J, Visotcky A, Braun N, Kerschner J, Tarima S, Brown D. Fiberoptic Endoscopic Evaluation of Swallowing in children: feeding outcomes related to diagnostic groups and endoscopic findings. Int J Pediatr Otorhinolaryngol. 2011 Aug;75(8):1024-31. doi: 10.1016/j.ijporl.2011.05.010. Epub 2011 Jun 12. PMID 21663978
- [Result] Dodrill P, Gosa MM. Pediatric Dysphagia: Physiology, Assessment, and Management. Ann Nutr Metab. 2015;66 Suppl 5:24-31. doi: 10.1159/000381372. Epub 2015 Jul 24. PMID 26226994